CLINICAL TRIAL: NCT05058014
Title: The International Skeletal Metastasis Registry
Brief Title: Skeletal Metastasis Registry
Status: Terminated | Type: Observational
Why Stopped: The original investigator, Dr. Forsberg moved to MSKCC and plan to open the study there.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Murtha Cancer Center (Unknown); Defense Health Programs with the U.S. Army Medical Research and Materiel Command (Unknown)
Responsible Party: Sponsor
Other Study IDs: SIB1802; IRB00157231 (Other: Johns Hopkins Medicine)
Record Dates: First submitted 2021-08-06; First posted 2021-09-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Bone Tumor
Keywords: Biopsy-proven or clinically-obvious metastatic bone disease
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational study designed to contribute data from patients with symptomatic metastatic bone disease treated at Sibley Memorial Hospital and Johns Hopkins Medicine to an international registry hosted by the Swedish Regional Cancer Centrum in Stockholm, Sweden. This protocol supports a worldwide effort to collect and store information from patients treated for symptomatic bone metastases within the International Skeletal Metastasis Registry (ISMR)

DETAILED DESCRIPTION:
The registry is designed to update a suite of clinical decision-support tools designed for use when treating patients with metastatic bone disease. The models estimate the likelihood of survival at 1, 3, 6, 12, 18, and 24 months post surgery, which in turn, may be used for surgical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 22 or older
* Biopsy-proven or clinically-obvious metastatic bone disease
* Symptomatic bone lesion requiring intervention o Including, not limited to, radiotherapy, cryotherapy, radiofrequency ablation, operative fixation, prosthetic replacement, amputation, or any combination of the above.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic bone disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 24 Months post surgery
  OS (in months) calculated from the date of intervention.

SECONDARY OUTCOMES:
Reoperation or retreatment for any reason | Up to 24 24 months post surgery
  Number of participants with reoperation or retreatment for any reason.
Time to reoperation or retreatment for any reason | Up to 24 months post surgery
  Timing of reoperation calculated from the date of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Levin, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States